CLINICAL TRIAL: NCT07373509
Title: Effectiveness of the Traumatic Brain Injury Whole Blood Test on Improving Assessment and Triage for Patients With GCS 13-15 Presenting to Emergency Departments
Brief Title: Emergency Department Implementation of the i-STAT Alinity Traumatic Brain Injury Whole Blood Test
Acronym: EDI
Status: Recruiting | Type: Observational
Sponsor: Shawn Eagle (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Shawn Eagle, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: STUDY25010137; HT94252510275 (Other Grant/Funding Number: Department of Defense; Dept. of the Army -- USAMRAA)
Record Dates: First submitted 2025-12-05; First posted 2026-01-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: TBI (Traumatic Brain Injury); Implementation Research
Keywords: Concussion; Traumatic Brain Injury; CT scan; Blood Biomarker; i-STAT Alinity TBI Test
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- ED Providers: Treating providers in the emergency department
- ED patients: Patients in the emergency department with GCS 13-15 with suspected TBI
  Interventions: Device: i-STAT Alinity TBI test

INTERVENTIONS:
Device: i-STAT Alinity TBI test — The i-STAT TBI cartridge is a point-of-care test that measures the level of biomarkers associated with brain injury in whole blood to help assess patients with suspected mTBI within 24 hours after injury.
  Groups: ED patients

SUMMARY:
The objective of this study is to identify determinants for implementing the i-STAT Alinity whole blood traumatic brain injury (TBI) test for its Food and Drug Administration (FDA)-indicated use and to evaluate other potential outcomes with clinical implications. The main questions it aims to answer are:

1. Determine the number of patients with non-elevated (i.e., below clinical cutoff) whole blood iSTAT Alinity tests who also receive CT scans.
2. What are the obstacles for using the i-STAT Alinity for its FDA-indicated use

DETAILED DESCRIPTION:
Objective:

The objective of this study is to utilize the integrated Promoting Action on Research Implementation in Health Services (i-PARIHS) framework to identify determinants for implementing the whole blood traumatic brain injury (TBI) test for its Food and Drug Administration (FDA)-indicated use and to evaluate other potential outcomes with clinical implications.

Specific Aims & working hypotheses:

Aim 1) Evaluate the effectiveness of the whole blood iSTAT Alinity test in determining the need for a head computed tomography (CT) scan in approximately 140 patients with a Glasgow Coma Score (GCS) 13-15 in the emergency department (ED) (approximately 47 per site) while assessing two novel outcomes with significant clinical implications (i.e., reduction in ED length of stay and predictive utility for ED revisits for the same injury).

• The working hypotheses are that the rate of patients with non-elevated (i.e., below clinical cutoff) whole blood iSTAT Alinity tests who also receive CT scans will mirror the preliminary study results (21 percent), a reduction in ED length of stay will be observed (in comparison to also receiving a CT scan) of greater than 3 hours, and predictive utility for return ED visits from the same injury will be high (area under the curve greater than 0.80).

Aim 2) Evaluate determinants for routine use of the whole blood iSTAT Alinity test by assessing acceptability, adoption, appropriateness and feasibility of the test at the organizational- and physician-level for each site and determine how these factors interplay with patient perspectives and knowledge to influence implementation of the test.

• The working hypotheses are that organization-, physician-, and patient-level determinants will be identified and gaps in patient knowledge will be observed. A diverse Community Advisory Board (CAB) will be assembled to provide important context of how these varying perspectives impact the whole blood iSTAT Alinity test utilization. We will also obtain community knowledge and perspective on this test via the CAB.

Aim 3) Develop a site-specific implementation blueprint for use of the whole blood iSTAT Alinity test in determining the need for a head CT scan and pilot test the blueprint in approximately 140 patients with GCS 13-15 in the ED (approximately 47 per site).

• The working hypothesis is that an implementation blueprint that targets identified determinants in Aim 2 will lead to a reduction in the rate of patients with negative whole blood iSTAT tests who also receive CT scan to 5 percent or less.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or older
2. Presenting to an enrolling ED with ED Arrival GCS of 13-15 following reported head blunt impact within 24 hours of injury
3. Meets Department of Defense (DoD) definition of mTBI:

A traumatically induced physiological disruption of brain function as a result of an external force that is indicated by new onset or worsening of at least one of the following clinical signs immediately following the event:

1. Any alteration of mental status (e.g., feeling dazed, disoriented, or confused)
2. Any period of loss of or a decreased level of consciousness, observed or self-report (loss of consciousness 30 minutes or less, an alteration of consciousness up to 24 hours)
3. Any loss of memory for events immediately before or after the injury (post-traumatic amnesia up to 1-day post-injury)

Exclusion Criteria:

1. Treating emergency department provider does not think a head CT scan is needed
2. Inability to obtain results for iSTAT Alinity TBI test within 24 hours of injury
3. Treating emergency department attending physician is not willing to participate
4. Pre-existing neurologic condition
5. Contraindication or inability to complete blood draw
6. Significant polytrauma that, in the opinion of the principal investigators, could impact peripheral GFAP levels or require a full body scan
7. History of penetrating TBI
8. History of neurosurgical intervention for previous TBI
9. Penetrating TBI for current injury
10. Any history of brain surgery
11. Any history of brain tumor
12. Patients on psychiatric hold

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency department providers and patients with suspected TBI
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Rate of CT scans completed | Up to 5 hours (from enrollment to CT scan completion)
  Rate of CTs completed for ED patient participants with a non-elevated i-STAT Alinity whole blood TBI test result.

SECONDARY OUTCOMES:
ED patient length of stay | Up to 5 hours (from arrival to discharge)
Patient return visit to ED | Up to two weeks
  Return visit for same injury within 2 weeks of initial visit
Military Acute Concussion Evaluation-2 (MACE-2) | Visit 1 (ED visit)
  MACE 2 is a 15-minute multimodal tool that assists providers in the assessment and diagnosis of concussion. It includes:
  1. An unscored screening section collected by clinician interview
  2. A cognitive exam with scores ranging 0-30; with higher scores representing better performance. A score of 25 or less is considered abnormal.
  3. Normal/Abnormal ratings of neurological function, symptom report, and visual-ocular functioning
  A total score is not generated.
Neurobehavioral Symptom Inventory (NSI) | The NSI will be completed once during the patient's visit 1 (ED visit), and once at visit 2 (2-week remote follow-up)
  The NSI is a 22-item scale of TBI symptoms which takes 2 minutes to complete. Total scores range from 0-88, with higher scores indicating more severe symptom burden.
Modified Rosenbaum Concussion Knowledge and Attitudes Survey (RoCKAS) | Visit 1 (ED visit)
  This is a 13-item survey to evaluate existing knowledge of concussion, which takes 2 minutes to complete. All questions are true/false. Correct responses get one point, with total scores ranging 0-13; higher scores indicate greater knowledge.
Mobilizing Implementation of iPARIHS Facilitation Planning Tool (Mi-PARIHS) | Visit 1 (enrollment) and again at 39 months (study conclusion)
  This is a 34-item survey to be filled out by ED providers to identify determinants for implementation of the I-STAT TBI test. Each item is rated with a 5-item likert-scale, rated -2 to +2, to identify barriers and facilitators/enablers for the i-STAT TBI test. Lower scores indicate more barriers.
Decisional Conflict Scale (DCS) | Visit 1 (enrollment) and again at 39 months (study conclusion)
  The DCS is a 16-item survey about decision-making to be filled out by ED providers. It measures 5 dimensions of decision making, with factors related to feeling uncertain, uninformed, unclear about values, unsupported, or ineffective decision making. All items are scored on a Likert scale ranging from 1 (strongly agree) to 5 (strongly disagree). Total scores range from 16-80; a higher score indicates a higher level of decisional conflict.
Implementation Questionnaire | Visit 1 (enrollment) and again at 39 months (study conclusion)
  This is a 4-item survey about the i-STAT TBI test implementation to be filled out by ED providers. All items are scored on a Likert scale ranging from 1 (completely disagree) to 5 (completely agree). Total scores range from 4-20; a higher score indicates a higher level of i-STAT TBI test implementation acceptance.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Eagle, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available through the Federal Interagency TBI Research
Time Frame: Shared scientific data will be made accessible as soon as possible, and no later than the time of an associated publication, or the end of performance period, whichever comes first.
Access Criteria: FITBIR qualified investigators will be provided access
URL: https://fitbir.nih.gov/